CLINICAL TRIAL: NCT05580523
Title: Aspirin Versus Metformin in Pregnancies at High Risk of Preterm Preeclampsia: a 3-arm Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Obstetrics & Gynecology Hospital of Fudan University (Other); Shanghai First Maternity and Infant Hospital (Other); West China Second University Hospital (Other); Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Chiu Yee Liona Poon, Professor (Clinical), Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MOST-AVERT
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Preeclampsia
Keywords: Preterm preeclampsia; Aspirin; Metformin
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: PI, participating research doctors, pharmacists at the local clinical trial pharmacy, project managers and others involved in the trial are all blinded to the investigational medicinal product (IMP). The tablets and capsules will be identical, so it will not be possible to distinguish between the different IMPs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aspirin 75 mg and placebo (Experimental): A capsule of 75 mg aspirin plus an aspirin identical-appearing capsule of placebo to be taken orally once per night from enrolment until 36 weeks' gestation and metformin identical-appearing placebo capsules to be taken orally twice per day from enrolment until delivery.
  Interventions: Drug: 75 mg acetylsalicylic acid; Drug: Placebo of acetylsalicylic acid and Metformin
- Aspirin 150 mg and placebo (Experimental): Two capsules of 75 mg aspirin to be taken orally once per night from enrolment until 36 weeks' gestation and metformin identical-appearing placebo capsules to be taken orally twice per day from enrolment until delivery.
  Interventions: Drug: 150 mg acetylsalicylic acid; Drug: Placebo of acetylsalicylic acid and Metformin
- Aspirin 75 mg and Metformin 1.5 g (Experimental): A capsule of 75 mg aspirin plus an aspirin identical-appearing capsule of placebo to be taken orally once per night from enrolment until 36 weeks' gestation and metformin capsules (up to 750 mg) to be taken twice per day from enrolment until delivery
  Interventions: Drug: 75 mg acetylsalicylic acid; Drug: 1.5g Metformin

INTERVENTIONS:
Drug: 75 mg acetylsalicylic acid — 75 mg acetylsalicylic acid (C9H8O4, CAS number 50-78-2) daily, Oral
  Other Names: 75mg Aspirin
  Arms: Aspirin 75 mg and Metformin 1.5 g; Aspirin 75 mg and placebo
Drug: 1.5g Metformin — up to 1.5 g metformin (C4H11N5, CAS number 657-24-9) daily, Oral Dose increases from 0.5g to 1.0g to 1.5g
  Other Names: 1.5g Glucophage
  Arms: Aspirin 75 mg and Metformin 1.5 g
Drug: 150 mg acetylsalicylic acid — 150 mg acetylsalicylic acid (C9H8O4, CAS number 50-78-2) daily, Oral
  Other Names: 150mg Aspirin
  Arms: Aspirin 150 mg and placebo
Drug: Placebo of acetylsalicylic acid and Metformin — Pills with shape, color and smell same with acetylsalicylic acid and metformin, daily, oral
  Arms: Aspirin 150 mg and placebo; Aspirin 75 mg and placebo

SUMMARY:
This is a prospective, multicenter, randomized controlled, double-blind trial of three treatment arms: (1) aspirin 75 mg/day vs. (2) aspirin 150 mg/day vs. (3) aspirin 75 mg/day with metformin 1.5 g/day from the first trimester to compare the incidence of preterm preeclampsia with delivery at <37 week's gestation between the treatment arms, in order to determine the optimal therapeutic intervention for the prevention of preterm preeclampsia among Chinese women at high-risk of preeclampsia.

DETAILED DESCRIPTION:
All women with singleton pregnancies who are attending for their routine hospital visit at 11-13 weeks' gestation will be invited to undergo screening for preeclampsia. We use a Bayes theorem-based method that combines maternal characteristics, medical and obstetric history together with mean arterial pressure (MAP) and serum placental growth factor (PlGF) level. Women who are deemed high-risk following first trimester combined screening (cutoff corresponding to a screen positive rate of 10%, e.g ≥1 in 80) will be invited to participate in the 3-arm randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies
* Live fetus at 11-13 weeks' gestation
* High-risk for preterm preeclampsia at 11-13 weeks by the algorithm combining maternal characteristics, medical and obstetric history, MAP and serum PlGF
* Informed and written consent

Exclusion Criteria:

* Age <18 years old
* Multiple pregnancies
* Treatment with low-dose aspirin and metformin at the time of screening
* Pregnancies complicated by major fetal abnormality identified during the first trimester
* Women with learning difficulties, or serious mental illness
* Bleeding disorders such as Von Willebrand's disease
* Active peptic ulceration or gastrointestinal bleeding
* Hypersensitivity to aspirin, metformin hydrochloride and other biguanides
* Treatment with long term nonsteroidal anti-inflammatory medication
* Hyperemesis gravidarum
* Renal, liver or heart failure
* A serious medical condition
* Concurrent participation in another drug trial or at any time within the previous 28 days
* Any other reason the clinical investigators think will prevent the potential participant from complying with the trial protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All eligible women with singleton pregnancies
Enrollment: 3000 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of preterm preeclampsia(<37 weeks) | ≥20 weeks to <37 weeks of gestation
  Preeclampsia will be defined as per the International Society for the Study of Hypertension in Pregnancy.The Proportions of delivery with preterm-preeclampsia between different intervention groups will be measured.

SECONDARY OUTCOMES:
Adverse outcome of pregnancy at <37 weeks. | <37 weeks of gestation
  including preeclampsia requiring delivery, gestational age (SGA; <5th percentile) requiring delivery, miscarriage or still birth or placental abruption.
Adverse outcome of pregnancy at <34 weeks. | <34 weeks of gestation
  including preeclampsia requiring delivery, gestational age (SGA; <5th percentile) requiring delivery, miscarriage or still birth or placental abruption.
Adverse outcome of pregnancy at ≥37 weeks | ≥37 weeks of gestation
  including preeclampsia requiring delivery, gestational age (SGA; <5th percentile) requiring delivery, stillbirth or placental abruption.
Neonatal mortality | During the first 28 days of life (0-27days)
  A neonatal death is a death during 0-27 days of life.
Neonatal morbidity | During the first 28 days of life (0-27days)
  Composite neonatal morbidity (any one of the following): >grade II intra-ventricular hemorrhage; neonatal sepsis confirmed by cultures; neonatal anemia requiring transfusion; respiratory distress syndrome requiring surfactant and ventilation; necrotising enterocolitis requiring surgical intervention.
Neonatal birthweight below the 3rd,5th and 10th centile. | At delivery
  Birthweight and birthweight percentile for gestational age at delivery is calculated using a normal range derived in a Chinese population.
Stillbirth or neonatal death | At delivery
  Stillbirth: the death of a baby before or during birth after 24 weeks of gestation. Neonatal death: the death of a baby within the first 28 days of life.
<34 weeks and <37 weeks spontaneous preterm delivery | At spontaneous delivery
  Spontaneous delivery at <34 weeks(early preterm) and at <37 weeks(total preterm) includes those with spontaneous onset of labor and those with preterm pre-labor rupture of membranes (PPROM).
Gestational age | At delivery
  Gestation is the period of time between conception and birth. During this time, the baby grows and develops inside the mother's womb. Gestational age is the common term used during pregnancy to describe how far along the pregnancy is. It is measured in weeks, from the first day of the woman's last menstrual cycle to the current date. A normal pregnancy can range from 38 to 42 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Chiu Yee, Liona Poon, MD, Principal Investigator — Chinese University of Hong Kong
Locations (6):
- China (6):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan

REFERENCES:
- [Background] Women's Heart Health Group of Chinese Society of Cardiology of Chinese Medical Association; Hypertension Group of Chinese Society of Cardiology of Chinese Medical Association. [Expert consensus on blood pressure management in hypertensive disorders of pregnancy (2019)]. Zhonghua Xin Xue Guan Bing Za Zhi. 2020 Mar 24;48(3):195-204. doi: 10.3760/cma.j.cn112148-20191024-00652. Chinese. PMID 32234176
- [Background] Witlin AG, Saade GR, Mattar F, Sibai BM. Predictors of neonatal outcome in women with severe preeclampsia or eclampsia between 24 and 33 weeks' gestation. Am J Obstet Gynecol. 2000 Mar;182(3):607-11. doi: 10.1067/mob.2000.104224. PMID 10739516
- [Background] Irgens HU, Reisaeter L, Irgens LM, Lie RT. Long term mortality of mothers and fathers after pre-eclampsia: population based cohort study. BMJ. 2001 Nov 24;323(7323):1213-7. doi: 10.1136/bmj.323.7323.1213. PMID 11719411
- [Background] von Dadelszen P, Magee LA, Roberts JM. Subclassification of preeclampsia. Hypertens Pregnancy. 2003;22(2):143-8. doi: 10.1081/PRG-120021060. PMID 12908998
- [Background] Chaemsaithong P, Pooh RK, Zheng M, Ma R, Chaiyasit N, Tokunaka M, Shaw SW, Seshadri S, Choolani M, Wataganara T, Yeo GSH, Wright A, Leung WC, Sekizawa A, Hu Y, Naruse K, Saito S, Sahota D, Leung TY, Poon LC. Prospective evaluation of screening performance of first-trimester prediction models for preterm preeclampsia in an Asian population. Am J Obstet Gynecol. 2019 Dec;221(6):650.e1-650.e16. doi: 10.1016/j.ajog.2019.09.041. Epub 2019 Oct 4. PMID 31589866
- [Background] Akolekar R, Syngelaki A, Sarquis R, Zvanca M, Nicolaides KH. Prediction of early, intermediate and late pre-eclampsia from maternal factors, biophysical and biochemical markers at 11-13 weeks. Prenat Diagn. 2011 Jan;31(1):66-74. doi: 10.1002/pd.2660. PMID 21210481
- [Background] Askie LM, Duley L, Henderson-Smart DJ, Stewart LA; PARIS Collaborative Group. Antiplatelet agents for prevention of pre-eclampsia: a meta-analysis of individual patient data. Lancet. 2007 May 26;369(9575):1791-1798. doi: 10.1016/S0140-6736(07)60712-0. PMID 17512048
- [Background] Rolnik DL, Wright D, Poon LC, O'Gorman N, Syngelaki A, de Paco Matallana C, Akolekar R, Cicero S, Janga D, Singh M, Molina FS, Persico N, Jani JC, Plasencia W, Papaioannou G, Tenenbaum-Gavish K, Meiri H, Gizurarson S, Maclagan K, Nicolaides KH. Aspirin versus Placebo in Pregnancies at High Risk for Preterm Preeclampsia. N Engl J Med. 2017 Aug 17;377(7):613-622. doi: 10.1056/NEJMoa1704559. Epub 2017 Jun 28. PMID 28657417
- [Background] Bujold E, Roberge S, Lacasse Y, Bureau M, Audibert F, Marcoux S, Forest JC, Giguere Y. Prevention of preeclampsia and intrauterine growth restriction with aspirin started in early pregnancy: a meta-analysis. Obstet Gynecol. 2010 Aug;116(2 Pt 1):402-414. doi: 10.1097/AOG.0b013e3181e9322a. PMID 20664402
- [Background] Roberge S, Villa P, Nicolaides K, Giguere Y, Vainio M, Bakthi A, Ebrashy A, Bujold E. Early administration of low-dose aspirin for the prevention of preterm and term preeclampsia: a systematic review and meta-analysis. Fetal Diagn Ther. 2012;31(3):141-6. doi: 10.1159/000336662. Epub 2012 Mar 21. PMID 22441437
- [Background] Roberge S, Nicolaides K, Demers S, Hyett J, Chaillet N, Bujold E. The role of aspirin dose on the prevention of preeclampsia and fetal growth restriction: systematic review and meta-analysis. Am J Obstet Gynecol. 2017 Feb;216(2):110-120.e6. doi: 10.1016/j.ajog.2016.09.076. Epub 2016 Sep 15. PMID 27640943
- [Background] Caron N, Rivard GE, Michon N, Morin F, Pilon D, Moutquin JM, Rey E. Low-dose ASA response using the PFA-100 in women with high-risk pregnancy. J Obstet Gynaecol Can. 2009 Nov;31(11):1022-1027. doi: 10.1016/S1701-2163(16)34346-8. PMID 20175340
- [Background] Rey E, Rivard GE. Is testing for aspirin response worthwhile in high-risk pregnancy? Eur J Obstet Gynecol Reprod Biol. 2011 Jul;157(1):38-42. doi: 10.1016/j.ejogrb.2011.02.026. Epub 2011 Mar 25. PMID 21440360
- [Background] Hypertensive Disorders in Pregnancy Subgroup, Chinese Society of Obstetrics and Gynecology, Chinese Medical Association. [Diagnosis and treatment of hypertension and pre-eclampsia in pregnancy: a clinical practice guideline in China（2020）]. Zhonghua Fu Chan Ke Za Zhi. 2020 Apr 25;55(4):227-238. doi: 10.3760/cma.j.cn112141-20200114-00039. Chinese. PMID 32375429
- [Background] Brownfoot FC, Hastie R, Hannan NJ, Cannon P, Tuohey L, Parry LJ, Senadheera S, Illanes SE, Kaitu'u-Lino TJ, Tong S. Metformin as a prevention and treatment for preeclampsia: effects on soluble fms-like tyrosine kinase 1 and soluble endoglin secretion and endothelial dysfunction. Am J Obstet Gynecol. 2016 Mar;214(3):356.e1-356.e15. doi: 10.1016/j.ajog.2015.12.019. Epub 2015 Dec 22. PMID 26721779
- [Background] Syngelaki A, Nicolaides KH, Balani J, Hyer S, Akolekar R, Kotecha R, Pastides A, Shehata H. Metformin versus Placebo in Obese Pregnant Women without Diabetes Mellitus. N Engl J Med. 2016 Feb 4;374(5):434-43. doi: 10.1056/NEJMoa1509819. PMID 26840133
- [Background] Chiswick C, Reynolds RM, Denison F, Drake AJ, Forbes S, Newby DE, Walker BR, Quenby S, Wray S, Weeks A, Lashen H, Rodriguez A, Murray G, Whyte S, Norman JE. Effect of metformin on maternal and fetal outcomes in obese pregnant women (EMPOWaR): a randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2015 Oct;3(10):778-86. doi: 10.1016/S2213-8587(15)00219-3. Epub 2015 Jul 9. PMID 26165398
- [Background] ACOG Practice Bulletin No. 202: Gestational Hypertension and Preeclampsia. Obstet Gynecol. 2019 Jan;133(1):1. doi: 10.1097/AOG.0000000000003018. PMID 30575675
- [Background] Poon LC, Volpe N, Muto B, Syngelaki A, Nicolaides KH. Birthweight with gestation and maternal characteristics in live births and stillbirths. Fetal Diagn Ther. 2012;32(3):156-65. doi: 10.1159/000338655. Epub 2012 Jul 26. PMID 22846512
- [Background] Wright D, Poon LC, Rolnik DL, Syngelaki A, Delgado JL, Vojtassakova D, de Alvarado M, Kapeti E, Rehal A, Pazos A, Carbone IF, Dutemeyer V, Plasencia W, Papantoniou N, Nicolaides KH. Aspirin for Evidence-Based Preeclampsia Prevention trial: influence of compliance on beneficial effect of aspirin in prevention of preterm preeclampsia. Am J Obstet Gynecol. 2017 Dec;217(6):685.e1-685.e5. doi: 10.1016/j.ajog.2017.08.110. Epub 2017 Sep 6. PMID 28888591
- [Derived] Liu J, Shen L, Nguyen-Hoang L, Zhou Q, Wang CC, Lu X, Sahota D, Chong KC, Ying H, Gu W, Zhou R, Yang H, Jiang Y, Chen D, Li X, Poon L. Aspirin versus metformin in pregnancies at high risk of preterm pre-eclampsia in China (AVERT): protocol for a multicentre, double-blind, 3-arm randomised controlled trial. BMJ Open. 2024 Apr 17;14(4):e074493. doi: 10.1136/bmjopen-2023-074493. PMID 38631826